CLINICAL TRIAL: NCT04200989
Title: Intra-lymphatic Immunotherapy for the Management of Peanut Allergy
Brief Title: Novel Treatment for Patients With Peanut Allergy: Intralymphatic Immunotherapy
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Scripps Health (Other)
Collaborators: The Scripps Research Institute (Other)
Responsible Party: Principal Investigator, Ronald A Simon, Emeritus Head, Division of Asthma, Allergy and Immunology, Scripps Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-19-7380
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2021-02

CONDITIONS: Food Allergy Peanut
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Intervention Model Description: All subjects receive the study intervention: Peanut ILIT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Peanut ILIT
  Interventions: Biological: Peanut allergen

INTERVENTIONS:
Biological: Peanut allergen — Intralymphatic immunotherapy injections.

SUMMARY:
Use of three intralymphatic injections of peanut allergen one month apart to induce tolerance to peanut in peanut allergic people.

DETAILED DESCRIPTION:
Eligible subject undergo a baseline blinded oral peanut challenge. Then the peanut ILIT as described above. Pretreatment with antihistamines, leukotriene modifier and albuterol before each treatment.

Following the three ILIT peanut injections a repeat blinded oral peanut challenge is performed.

Blood is drawn at each of the 5 study visits for a variety of tests trying to elucidate the mechanism(s) of the induction of tolerance to peanut.

ELIGIBILITY:
Inclusion Criteria:

History of peanut allergy Positive prick skin tests or invitro IgE to peanut Positive blinded oral peanut challenge.

-

Exclusion Criteria:

History of

* life threatening anaphylaxis to peanut Uncontrolled asthma

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Peanut tolerance | 4 months
  Increase in amount (mg - grams) of peanut ingested without reaction from baseline to one month post ILIT

CONTACTS AND LOCATIONS:
Overall Officials: Simon A Ronald, MD, Principal Investigator — Scripps Health
Locations (1):
- Scripps Clinic, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Senti G, Crameri R, Kuster D, Johansen P, Martinez-Gomez JM, Graf N, Steiner M, Hothorn LA, Gronlund H, Tivig C, Zaleska A, Soyer O, van Hage M, Akdis CA, Akdis M, Rose H, Kundig TM. Intralymphatic immunotherapy for cat allergy induces tolerance after only 3 injections. J Allergy Clin Immunol. 2012 May;129(5):1290-6. doi: 10.1016/j.jaci.2012.02.026. Epub 2012 Mar 30. PMID 22464647
- [Background] Hylander T, Latif L, Petersson-Westin U, Cardell LO. Intralymphatic allergen-specific immunotherapy: an effective and safe alternative treatment route for pollen-induced allergic rhinitis. J Allergy Clin Immunol. 2013 Feb;131(2):412-20. doi: 10.1016/j.jaci.2012.10.056. PMID 23374268
- [Background] Lee SP, Choi SJ, Joe E, Lee SM, Lee MW, Shim JW, Kim YJ, Kyung SY, Park JW, Jeong SH, Jung JH. A Pilot Study of Intralymphatic Immunotherapy for House Dust Mite, Cat, and Dog Allergies. Allergy Asthma Immunol Res. 2017 May;9(3):272-277. doi: 10.4168/aair.2017.9.3.272. PMID 28293934